CLINICAL TRIAL: NCT07203469
Title: Where Wild Things Grow: Immediate and Long-term Impact of Nature- and Activity-based Group Interventions for Neurodivergent Children and Youth in School, Health Care and Leisure Settings in Agder
Brief Title: Where Wild Things Grow: Nature- and Activity-based Group Interventions for Neurodivergent Children and Youth
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sorlandet Hospital HF (Other Government)
Collaborators: University of Agder (Other); University of Stavanger (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REC nr. 807380
Record Dates: First submitted 2025-09-16; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Neurodevelopmental Outcomes; ADHD - Attention Deficit Disorder With Hyperactivity; Autism; Tourette Syndrome; Health-Related Quality-of-Life; Heart Rate Variability (HRV)
Keywords: Nature-based; Action research; child and adolescent mental health; ADHD; Autism; Health-related quality of life; outdoor therapy; experiential education; heart rate variability
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Autistic Disorder; Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- School setting (PhD 1) (Active Comparator): In this study arm, we compare two approaches to nature-based experiential learning.
  Interventions: Behavioral: Universal approach; Behavioral: Selective approach
- Health Care Setting (PhD 2) (Active Comparator): In this study arm, we compare two nature- and activity-based group treatments.
  Interventions: Behavioral: Outdoor therapy; Behavioral: Climbing therapy
- Heart Rate Variability (Substudy 1) (Experimental): Heart rate variability (HRV) is measured across contexts to explore physiological outcomes and stress levels
  Interventions: Behavioral: Universal approach; Behavioral: Selective approach; Behavioral: Outdoor therapy; Behavioral: Climbing therapy

INTERVENTIONS:
Behavioral: Universal approach — In this intervention, the whole class participates in a 12-week nature-based experiential education program
  Other Names: Universell Friluftslæring
  Arms: Heart Rate Variability (Substudy 1); School setting (PhD 1)
Behavioral: Selective approach — In this intervention, an intentional group of pupils with an identified need is recruited from different classes within the same school to participate in a 12-week nature-based experiential education program
  Other Names: Selektiv Friluftslæring
  Arms: Heart Rate Variability (Substudy 1); School setting (PhD 1)
Behavioral: Outdoor therapy — This intervention is a 10-week outdoor therapy group treatment that takes place in nearby nature
  Other Names: Friluftsterapi; Basecamp
  Arms: Health Care Setting (PhD 2); Heart Rate Variability (Substudy 1)
Behavioral: Climbing therapy — This intervention is a 10-week climbing therapy group treatment that takes place indoors in a climbing hall
  Other Names: Klatreterapi
  Arms: Health Care Setting (PhD 2); Heart Rate Variability (Substudy 1)

SUMMARY:
The goal of this action research project is to develop and implement nature- and activity-based group interventions across health care, school and leisure settings in Southern Norway. The interventions are tailored to support the mental health, self-efficacy and daily life functioning of children and youth in the Agder region, with a particular focus on youngsters who struggle due to neurodivergence, such as Attention Deficit Hyperactivity Disorder (ADHD), Autism Spectrum Disorder (ASD) or Tourette's syndrome.

The main questions we aim to answer are:

1. To what extent does nature- and activity-based outdoor education contribute to improvements in children's quality of life?
2. To what extent does nature- and activity-based interventions in a health care setting improve children's self-efficacy, self-esteem and quality of life?
3. Is there a difference in physiological reactions between nature-based provision of education or therapy and traditional indoor provision of education or therapy?

Participants will take part in a 12-week school-based or health care intervention.

DETAILED DESCRIPTION:
BACKGROUND Today's children grow up in uncertain times. Global trends include the multicrisis of climate change, pandemic and wars, lack of contact with nature and a life supercharged with technology that offers unprecedented possibilities, but is simultaneously associated with loneliness and distress. Factors such as these may underlie the sharp decline in mental well-being in Norwegian youth during the previous two decades. Indeed, it has been noted that increased screen time is associated with increased depression and anxiety in Norwegian youth and further that replacing free, imaginative outdoor play with more time spent online is an important factor underlying the mental health crisis.

When it comes to neurodivergent population more specifically, numerous intertwined issues are especially pronounced for neurodiverse children and youth, who are at an increased risk of developing mood disorders, planning or committing suicide, becoming delinquent and misusing substances compared to their neurotypical peers.

These complex needs of neurodiverse children combined with the sharp rise in referrals to health services, call for proactive collaboration between schools, healthcare services, community-based services and interest organizations. Clinicians, researchers, politicians and the youth themselves have called for systemic and low-threshold interventions, preferably aimed at strengthening a positive self-image and personal resources, rather than concentrating on reduction of symptoms and deficits. One path forward is to develop tailored group interventions that foster individual inclusion and mastery, while being adaptable for regional implementation across a continuum of services. Over time, this process could ideally lead to systemic societal change by better nurturing the developmental needs of neurodiverse children and youth.

In Where Wild Things Grow, a collaborative continuum across educational, health care and leisure sectors has been established to build systemic competence and to develop, implement and test nature- and activity-based group interventions for neurodivergent children and youth. If effective, the interventions and the collaborative model can be replicated nationally and internationally in a systemic, joint effort to promoting children's overall growth, development and well-being.

The interventions are informed by the global trends outlined above, research on nature-based approaches for children with ADHD and autism, strength-based approaches and the neurodiversity movement. Studies have shown that outdoor education has positive effect on children's biological stress regulation and brain development and function, where children participating in outdoor schooling in a forest exhibited a healthier diurnal rhythm compared to those in a traditional school setting. Similarly, Dettweiler et al. demonstrated that outdoor education fosters better stress regulation and brain development, particularly in those areas of the brain that are associated with stress response and cognitive control. Furthermore, this project builds on a decade of clinical studies by a collective of researchers and practitioners at Sorlandet Hospital that has focused on developing transdiagnostic nature- and activity-based interventions for children, youth, and families.

In Where Wild Things Grow, we will develop and implement various nature- and activity-based group interventions, including two versions of nature-based outdoor education: (1) a universal approach (Universell Friluftslæring; UFL), which includes all pupils, and (2) a selective approach (Selektiv Friluftslæring; SFL), which includes an intentional selection of pupils with identified needs. In the health care setting, we implement: (3) an adapted version of outdoor therapy (Friluftsterapi; FT) that applies short microexpeditions in nearby nature, integrated with resource- and recovery-focused therapy, and (4) Climbing Therapy (Klatreterapi; KT), which combines group activities in an indoor climbing hall with techniques from Cognitive Behavioral Therapy (CBT). Finally, adapted versions of the abovementioned nature- and activity-based interventions will be offered as low-threshold, yet supportive, initiatives through interest organizations and municipal services in the Agder region as a follow-up activity in order to sustain positive development and community over time.

These interventions are intended to complement standard education and treatment, as well as ensure sustainability over time.

Neurodivergent youth often struggle with recognizing their bodily states and emotions and sustaining attention, which may cause distress in ordinary classroom education and talk-based therapy. By moving learning and therapeutic work into nature or climbing environments, nature- and activity-based interventions aim to engage participants more effectively. Integrating experiential learning and therapeutic practices with group exercises and physical movement creates a "natural laboratory" for exploring feelings, thoughts, and bodily reactions as they arise. Theoretically, our approach draws on Self-Determination Theory, Self-Efficacy Theory, Outdoor Therapy, Outdoor Education, the psychological, physiological and social benefits of nature contact and the CBT framework underlying therapeutic climbing. It is particularly informed by recent research on nature-based interventions to improve the quality of life of autistic children, including social interactions and adapting to change, as well as helping children with ADHD concentrate. Further, physical activity is an effective intervention in itself, recently shown to be on par with psychotherapy and pharmacological treatments.

Heart Rate Variability (HRV) is a measurable indicator of the autonomic nervous system's (ANS) regulation of the heart. HRV reflects the balance between the sympathetic nervous system (SNS), which activates the body's "fight or flight" response, and the parasympathetic nervous system (PNS), which promotes relaxation and recovery. HRV is a key metric for understanding physiological responses to stress. Stress involves mental strain or pressure that can arise from various tasks such as problem solving, decision-making, or coping with challenging situations. It activates the body's stress response systems, primarily involving the hypothalamic-pituitary-adrenal (HPA) axis and the ANS. During stressful tasks, stress often results in the withdrawal of parasympathetic (vagal) activity. The PNS is responsible for promoting relaxation and recovery. Reduced parasympathetic activity leads to less variability in the heart rate, contributing to lower HRV. HRV is also an indicator of social stress, which can occur in social interactions and group settings. Social stress activates similar physiological pathways as cognitive stress, involving the ANS and HPA axis. High social stress can lead to reduced HRV, indicating lower parasympathetic activity and higher sympathetic activation. This makes HRV a valuable measure for understanding how social environments, such as outdoor school or therapy activities may impact physiological stress responses.

HYPOTHESES, AIMS AND OBJECTIVES This project aims to investigate the immediate and long-term impact of nature- and activity-based group interventions for neurodiverse youth across school, health care and leisure settings, while identifying any contraindications to their use. It contributes to the debate on the efficacy of nature-based interventions for youth with ADHD, with some studies reporting strong effects and others none. It also addresses the mixed findings on the impact of nature contact on the well-being, emotional regulation and social relationships of autistic youth, with some studies showing positive effects, and others negative ones. More specifically, the various studies will explore the immediate impact on physiological reactions across intervention and ordinary settings in school and health care contexts, and the immediate and long-term impact of the interventions on the self-esteem, self-efficacy and quality of life of neurodiverse youth. Additionally, it aims to acquire greater insights into the preventative and health-promoting potential of multi-dimensional group interventions that combine cognitive, emotional, physical and social dimensions and that take place in non-school or non-clinical environments.

The project comprises two PhD-projects (PhD 1 in a school setting and PhD 2 in a health care setting), in addition to Substudy 1, which takes place in both school and health care settings. We explore the following research objectives and questions:

PhD 1:

I. How and why have teachers implemented nature-based outdoor education? The objective of PhD 1 is to operationalize various understandings of nature-based outdoor education in order to develop a preventative method that can be implemented across Agder schools in the main study.

II. How do teachers, parents and children perceive the impact of outdoor education on children's quality of life? The next objective is to explore the immediate impact of outdoor education on the pupils' quality of life from various perspectives.

III. To what extent does nature-based outdoor education contribute to improvements in children's quality of life over a school semester? And finally, exploring the longer-term impact of outdoor education.

PhD 2:

I. Impact of Interventions: To what extent does FT and CT improve children's self-efficacy, self-esteem, and quality of life compared to pre-intervention baselines? Are benefits sustained at follow-up measurements at 3, 6, and 12 months? II. What works for whom and under which circumstances in nature- and activity-based interventions? The second objective is to gain in-depth knowledge of how to best support the self-efficacy, self-esteem and quality of life of neurodiverse youth, and contraindications to its use.

Substudy 1:

I. Are there differences in physiological stress levels between outdoor and indoor provision of education and therapy? II. If outdoor provision of education and therapy leads to less physiological stress, can level of physical activity explain some of the variance in the data? The objective of Substudy 1 is to examine whether there is a difference in physiological reactions, measured by heart rate (HR) and heart rate variability (HRV), between outdoor and classroom teaching, and between outdoor and indoor provision of therapy. We aim to determine if the body reacts differently in nature compared to a traditional classroom or therapy setting, and whether physical activity levels can explain variance in data especially related to physiological stress.

PROJECT METHODOLOGY

Participants PhD 1: Participants are pupils who participate in nature- and activity-based outdoor education offered through participating schools. In the pilot phase, three schools participate in the development of the interventions. For the main study, fourteen additional schools will be recruited. The schools choose how many interventions they will facilitate during the project period.

PhD 2: Participants are children and adolescents aged 12-18 years of age that have been referred to specialist mental health care at ABUP at Sorlandet Hospital in Kristiansand or Arendal, or to municipal services in Agder. Exclusion criteria include substance misuse, acute psychosis, current suicidal behavior or ideation, and severe eating disorders. Medication is treated as a moderator variable rather than an inclusion or exclusion criterion, as the focus is on quality of life, self-esteem, and self-efficacy rather than neuropsychiatric symptoms.

Substudy 1: Participants are recruited from both PhD 1 and PhD 2. We aim to include a minimum of two interventions from the pilot schools, recruiting anywhere from 12- 16 pupils (n= 12- 16) aged 13- 15 years of age from WP 1. Next, we aim to include a minimum of one FL and one CL from Sørlandet sykehus, recruiting anywhere from 10- 14 youth (n= 10- 14) aged 12- 18 years of age from WP 2.

During the autumn of 2024 and spring of 2025, all interventions underwent a pilot phase, during which all the interventions were implemented according to the manuals, upon necessary adjustments were made and data collection methods and practical arrangements tested, in preparation for the main study phase commencing i September 2025.

Quantitative and qualitative methods PhD 1: One questionnaire will be utilized in this substudy, where the KIDSCREEN-27 (KIDS) will be applied to investigate the extent to which nature-based outdoor education contributes to the improvements of children's quality of life. KIDSCREEN-27 is a validated instrument designed to assess health-related quality of life in children and adolescents across various dimensions, including physical and psychological well-being, social relationships and the school environment.

PhD 2: Quality of life functions as the main outcome measure. It is operationalized as single items related to happiness (SIHa), health (SIHe), stress (SIS) and the dimensions of well-being operationalized in an Outcome Rating Scale, together with KIDSCREEN-10 (KIDS). Secondary outcomes (exploratory analyses) are Goal-based outcome (GBO), Mental Health Promoting Knowledge, Rosenberg Self-esteem Scale (RSES) and the Behaviours and Feelings Survey (BFS). At the end of each session, we collect a Group Session Rating Scale. In addition, we collect KIDSCREEN-10 and BRIEF-2 from parents and the Strength- and Difficulties Questionnaire (SDQ) and BRIEF-2 from teachers, in addition to monitoring school absence.

Data analysis is based on the multiple baseline design (MBD), a single-case experimental approach well-suited to the project's action research focus. In MBD, each participant serves as their own control with varying baseline lengths, allowing for systematic observation of changes and helping establish causality by showing changes occur post-intervention rather than due to other factors.

To explore the educational and therapeutic opportunities for neurodivergent children in non-school and non-clinical environments like nature or climbing halls, we apply the constructivist grounded theory methodology to build empirically and clinically relevant insights and knowledge that can improve the precision and impact of outdoor education and mental health treatment for neurodivergent populations. Data collection includes participant observation and individual interviews alongside quantitative measurements, continuing until theoretical saturation, thus achieving a comprehensive description and conceptualization of the educational and health-promoting potentials and hindrances of group-based out-door education and therapy for neurodiverse populations.

Predicting participant recruitment and retention in youth clinical research is challenging. However, using multiple baseline and grounded theory data collection ensures an in-depth exploration of neurodiverse populations' needs and the educational and health-promoting impact of interventions, regardless of sample size. This scalable design, from a single case to multiple participants, guarantees study completion, with the multiple baselines approach enabling effective use of quantitative data even if challenges arise.

Substudy 1: Wearable devices (e.g., Polar H10 heart rate sensor) provide a non-invasive way to measure HRV and physical activity via accelerometry, offering insights into the physiological responses of students in the different learning environments. Key HRV metrics include: Heart Rate (HR): The number of heart-beats per minute. Higher HR can indicate increased activation or arousal. Root Mean Square of Successive Differences (RMSSD): An HRV metric that measures short-term variations in heartbeats. Reduced RMSSD can indicate decreased parasympathetic activity and increased stress. Percentage of successive R-R inter-vals that differ by more than 50 ms (pNN50): Another HRV metric reflecting parasympathetic activity. Reduced pNN50 can indicate increased stress. This quasi-experiment seeks to answer the research ques-tion if outdoor provision of education or therapy leads to less physiological stress, and if the level of phys-ical activity can explain some of the variance in the data.

Data from the heart rate monitors will be analyzed using Dynamic Structural Equation Modeling (DSEM) on the three above introduced HRV metrics, which will be calculated for epochs of 5 min for the duration of the respective teaching session. DSEM is an advanced statistical method that allows for the analysis of intensive longitudinal data and can model dynamic processes over time. This approach provides insights into intra-individual trajectories and between-individual differences in both contexts. Additionally, DSEM allows for the parallel modeling of physical activity and stress, enabling cross-lagged inferences about their relationship. Data from the questionnaire are included on the between-level as control variables.

PROJECT GROUP AND DISSEMINATION The project group comprises pedagogues, clinicians and researchers form Sorlandet Hospital, University of Agder and University of Agder, as well as four user representatives from local interest organizations, who will meet quarterly throughout the project period to address any potential dilemmas, including ethical and methodological concerns.

In addition to scientific publications, results will be disseminated at national and international conferences. Key achievements will be highlighted in periodic press releases throughout the project. Plans and results will be widely disseminated through various channels to health authorities, health personnel, patient groups, and scientific communities regionally, nationally and internationally. Local interest organizations (ADHD, Autism, Tourette's Associations and "En skole for alle") will communicate with their national counterparts. The project will conclude with a hybrid seminar in Norwegian in May 2028 and an online webinar in English in June 2028 to ensure broad dissemination of findings.

ELIGIBILITY:
Inclusion Criteria:

* In PhD 1, participants are recruited on class-level (all) or individual (identified need).
* In PhD 2, inclusion criteria are patients that participate in the specific interventions.

Exclusion Criteria:

* In PhD 2, exclusion criteria include substance misuse, acute psychosis, current suicidal behavior/ideation, and severe eating disorders.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Quality of life (PhD 2) | Up to 12 months after a 10-week intervention
  Operationalized as single items on hapiness, health, stress, outcome rating scale and KIDSCREEN-10
Health-related quality of life (PhD 1) | Up to four weeks after a 12- week intervention
  Measured by KIDSCREEN-27
Physiological reactions | One day data collection during 12-week intervention. No follow-up.
  Measured by heart rate and heart rate variability

CONTACTS AND LOCATIONS:
Overall Officials: Carina R Fernee, PhD, Principal Investigator — Sørlandet Hospital HF
Locations (2):
- Norway (2):
  - Department of Child and Adolescent Mental Health (ABUP), Sørlandet Hospital HF, Kristiansand, Agder
  - Department of Sport and Physical Education, University of Agder, Kristiansand, Agder

IPD SHARING:
Plan to Share IPD: No
It is not planned to share IPD, but we will consider each individual request for data sharing.

REFERENCES:
- See also: This is a project website for Where Wild Things Grow, or "Vill Vekst" in Norwegian — https://www.uia.no/forskning/prosjekter/helse-idrett/vill-vekst/index.html